CLINICAL TRIAL: NCT04294225
Title: Pharmacodynamic Study of Estrogen Suppression Threshold-Directed Therapy (ESTDT) of Anastrozole as Adjuvant Therapy for Early Stage Breast Cancer
Brief Title: Anastrozole and Letrozole After Surgery for the Treatment of Stage I-III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1931; NCI-2020-01062 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1931 (Other: Mayo Clinic in Rochester); P30CA015083 (NIH); P50CA116201 (NIH)
Record Dates: First submitted 2020-02-26; First posted 2020-03-04 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2023-10

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Early-Stage Breast Carcinoma; Invasive Breast Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (anastrozole, letrozole) (Experimental): Patients receive anastrozole PO QD for 56-70 days (8-10 weeks). Patients with E1 >= 1.3 pg/ml and E2 >= 0.5 pg/ml continue to receive anastrozole PO QD for another 56-70 days (8-10 weeks). Patients then receive letrozole PO QD for 8-10 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anastrozole; Drug: Letrozole

INTERVENTIONS:
Drug: Anastrozole — Given PO
  Other Names: Anastrazole; Arimidex; ICI D1033; ICI-D1033; ZD-1033
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara

SUMMARY:
This phase II trial studies how well anastrozole and letrozole after surgery work in treating patients with stage I-III breast cancer. Drugs, such as anastrozole and letrozole, may stop the growth of tumor cells by decreasing the amount of estrogen made by the body. Giving anastrozole and letrozole after surgery may prevent breast cancer from coming back (recurrence).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the proportion of women who have adequate estrone (E1) and estradiol (E2) suppression after 8-10 weeks of adjuvant anastrozole 10 mg once daily (ANA10) having had inadequate E1 and E2 suppression after 8-10 weeks of standard dose anastrozole 1 mg once daily (ANA1).

SECONDARY OBJECTIVES:

I. To estimate the proportion of women with elevated E1 and E2 levels after 8-10 weeks of adjuvant ANA1.

II. To estimate the proportion of women with elevated E1 and E2 levels after 8-10 weeks of adjuvant ANA1 whose E1 and E2 levels remain elevated after 8-10 weeks of adjuvant ANA10.

III. To examine the toxicity profile of ANA1 over the 8-10 weeks of treatment, ANA10 over the 8-10 weeks of treatment, and letrozole over the 8-10 weeks of treatment.

IV. To examine concentrations of anastrozole at both the ANA1 and ANA10 dose levels.

V. To examine E1 and E2 concentrations, as well as letrozole drug levels, in patients receiving letrozole (following ANA10).

VI. To bank deoxyribonucleic acid (DNA) for examination of single-nucleotide polymorphism (SNP)-set(s) determined in the ongoing Mayo Clinic Breast Cancer Specialized Program of Research Excellence (SPORE) Project 4.

EXPLORATORY OBJECTIVE:

I. To examine association between clinical variables such as age, age at menopause, body mass index (BMI), receipt of chemotherapy, chemotherapy regimen, and dose on E1 and E2 levels after 8-10 weeks of ANA10.

OUTLINE:

Patients receive anastrozole orally (PO) once daily (QD) for 56-70 days (8-10 weeks). Patients with E1 >= 1.3 pg/ml and E2 >= 0.5 pg/ml continue to receive anastrozole PO QD for another 56-70 days (8-10 weeks). Patients then receive letrozole PO QD for 8-10 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION-INCLUSION CRITERIA
* Disease characteristics:

  * Histological confirmation of invasive breast carcinoma
  * Stage I-III breast cancer
  * Estrogen receptor (ER) positive disease according to American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines as ER >= 1% positive nuclear staining
* Completion of all planned cancer treatments prior to registration:

  * Surgical resection of breast and nodal surgery; (NOTE: Reconstructive surgery does not have to be completed)
  * Adjuvant radiation therapy, if needed
  * Neoadjuvant and/or adjuvant chemotherapy, if needed
* Post-menopausal defined as

  * Age >= 60 and amenorrhea > 12 consecutive months OR
  * Previous bilateral oophorectomy OR
  * Age < 60 and amenorrhea > 12 consecutive months and documented follicle stimulating hormone (FSH) level within post-menopausal range according to institutional standard

    * NOTE: Patients who did not meet these criteria at time of diagnosis and received pre-operative (neoadjuvant) or post-operative (adjuvant) chemotherapy will not be allowed to participate
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Hemoglobin >= 8.0 g/dL (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 70,000/mm^3 (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (obtained =< 14 days prior to registration)
* Ability to swallow oral medication
* Provide written informed consent
* Willingness to provide mandatory blood specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* RE-REGISTRATION-INCLUSION CRITERIA
* Confirmation that baseline blood sample was drawn and submitted
* Blood estrogen levels after cycle 1 anastrozole (ANA1) must meet the following criteria:

  * E1 >= 1.3 pg/ml, AND
  * E2 >= 0.5 pg/ml

Exclusion Criteria:

* REGISTRATION-EXCLUSION CRITERIA
* Pre-menopausal women receiving ovarian function suppression (goserelin, leuprolide, etc.)
* Stage IV (metastatic) breast cancer
* HER2 positive breast cancer as defined by

  * HER2 immunohistochemistry (IHC) >= 3+
  * HER2/CEP17 >= 2.0
  * HER2/CEP17 < 2.0 and average HER2 copy number of >= 6.0 signals/cell
* Prior endocrine therapy for this breast cancer. Exceptions:

  * Pre-operative aromatase therapy (anastrozole, letrozole, or exemestane) and last treatment was >= 4 weeks prior to registration OR
  * Pre-operative tamoxifen therapy and last treatment was >= 12 weeks prior to registration
* Currently receiving any of the following cancer-directed therapies:

  * Radiation therapy
  * Systemic therapy such as chemotherapy (standard or investigational)
* Bisphosphonate therapy started < 4 weeks prior to registration

  * NOTE: If patient is currently on bisphosphonate therapy she must be on stable dose for >= 4 weeks prior to registration. Patients not currently taking bisphosphonates will be allowed to start bisphosphonate therapy after completion of anastrozole (1 mg and 10 mg daily [if given]). Information regarding bisphosphonate therapy will be collected
* Current use of systemic or topical exogenous estrogen or progesterone (menopausal hormone replacement therapy [HRT])
* Prior ovarian function suppression (leuprolide, goserelin, etc.)
* Inability to provide informed consent
* History of contralateral ductal carcinoma in situ (DCIS) or invasive breast cancer

  * NOTE: Exception allowed if

    * Patient did not receive adjuvant endocrine therapy OR
    * Patient received adjuvant endocrine therapy but has been off treatment for at least 6 months prior to registration
* Concurrent active malignancy or history of malignancy =< 3 years prior to registration

  * NOTE: Exceptions allowed for successfully treated cervical carcinoma in situ, lobular carcinoma in situ of the breast, papillary thyroid cancer, or non-melanoma skin cancer
* Prior prevention therapy with an aromatase inhibitor or a selective estrogen receptor modulator (SERM). Exception: Therapy with a SERM (tamoxifen or raloxifene) is allowed if patient has been off treatment for >= 6 months prior to registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tufia C Haddad, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Anastrozole, Letrozole): Patients were to receive anastrozole 1 mg daily for 8 weeks (ANA1). After 8 weeks of ANA1, patients with E1 < 1.3 pg/ml and/or E2 < 0.5 pg/ml completed study and patients with E1 >= 1.3 pg/ml and E2 >= 0.5 pg/ml were to switch to anastrozole 10 mg daily (ANA10) for 8 weeks. After 8 weeks of ANA10, patients were to switch to letrozole 2.5 mg daily for 8 weeks. E1 and E2 levels were measured after this 8 week period. Patients were then go off study
Period: Anastrozole 1 mg/Day
Arm/Group | Treatment (Anastrozole, Letrozole)
Started | 158
Completed | 147
Not Completed | 11
Not completed — Discontinued due to COVID | 1
Not completed — Discontinued due to adverse events | 3
Not completed — Withdrawal by Subject | 5
Not completed — Ineligible | 2
Period: Anastrozole 10 mg/Day
Arm/Group | Treatment (Anastrozole, Letrozole)
Started | 33
Completed | 32
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Letrozole 2.5 mg/Day
Arm/Group | Treatment (Anastrozole, Letrozole)
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients that began treatment and are eligible are included in the analysis population
Arm/Group | Treatment (Anastrozole, Letrozole)
Number analyzed (Participants) | 156
Age, Customized [Count of Participants; unit: Participants]
  Age at registration (years): 40-49 | 5
  Age at registration (years): 50-59 | 46
  Age at registration (years): 60-69 | 62
  Age at registration (years): 70-79 | 35
  Age at registration (years): 80-89 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 149
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 146
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 156
BMI [Count of Participants; unit: Participants] — Underweight/Normal = (BMI<25.0)> Overweight = (25.0<=BMI<30.0)> Obese = (BMI>=30.0)
  Participants
    Underweight/Normal | 36
    Overweight | 54
    Obese | 62
    Unknown | 4
ECOG Performance Status [Count of Participants; unit: Participants] — 0 - Fully active, able to carry on all pre-disease performance without restriction; 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; 3 - Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; 4 - Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; 5 - Dead
  Participants
    0 | 148
    1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adequate Estrogen Suppression After 8 Weeks of Adjuvant Anastrozole 10 mg Daily
Description: Percentage of women who have adequate E1 and E2 suppression (E1 < 1.3 pg/ml and/or E2 < 0.5) after 8-10 weeks of adjuvant anastrozole 10 mg daily having had inadequate E1 and E2 (E1 >= 1.3 pg/ml and E2 >= 0.5) after 8-10 weeks of adjuvant anastrozole 1 mg daily.
Time Frame: 24 weeks
Population: Only participants that received anastrozole 10 mg daily (ANA10) and were adherent (reported taking ANA10 for 45-84 days) to treatment were analyzed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Anastrozole, Letrozole)
Number analyzed (Participants) | 25
percentage of participants | 76.0 [58.1 to 89.0]

2. Secondary Outcome: Number of Participants Experiencing a Grade 3 or Greater Adverse Event
Description: Patients will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Patients were to receive anastrozole 1 mg daily for 8 weeks (ANA1). After 8 weeks of ANA1, patients with E1 < 1.3 pg/ml and/or E2 < 0.5 pg/ml completed study and patients with E1 >= 1.3 pg/ml and E2 >= 0.5 pg/ml were to switch to anastrozole 10 mg daily (ANA10) for 8 weeks. After 8 weeks of ANA10, patients were to switch to letrozole 2.5 mg daily for 8 weeks. E1 and E2 levels were measured after this 8 week period. Patients were then go off study
Time Frame: 24 weeks
Population: Only participants that received treatment and were eligible were analyzed
Measure: Count of Participants; unit: Participants
Groups:
- Anastrozole 1mg Daily: Anastrozole 1mg daily
- Anastrozolem10mg Daily: Anastrozolem10mg daily
- Letrozole 2.5 mg Daily: Letrozole 2.5 mg Daily
Arm/Group | Anastrozole 1mg Daily | Anastrozolem10mg Daily | Letrozole 2.5 mg Daily
Number analyzed (Participants) | 156 | 33 | 24
Participants | 6 | 0 | 0

3. Secondary Outcome: Percent Change in Estrone (E1) and Estradiol (E2) Concentrations
Description: Descriptive statistics will be used. The median percent change in E1 and E2 concentrations from pre-AI levels will be presented.
Time Frame: 24 weeks
Population: Patients that received anastrozole 10 mg daily (ANA10) and were adherent to treatment were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Treatment (Anastrozole, Letrozole)
Number analyzed (Participants) | 25
percent change
  E1 levels | -97.0 [-98.1 to -95.0]
  E2 levels | -94.6 [-96.7 to -89.7]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Anastrozole 10mg Daily: Anastrozole 10mg daily
Arm/Group | Anastrozole 1mg Daily | Anastrozole 10mg Daily | Letrozole 2.5 mg Daily
All-Cause Mortality (participants affected / at risk) | 0/156 | 0/33 | 0/24
Serious Adverse Events (participants affected / at risk) | 4/156 | 1/33 | 0/24
Other Adverse Events (participants affected / at risk) | 120/156 | 26/33 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anastrozole 1mg Daily (N=156) | Anastrozole 10mg Daily (N=33) | Letrozole 2.5 mg Daily (N=24)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Breast infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anastrozole 1mg Daily (N=156) | Anastrozole 10mg Daily (N=33) | Letrozole 2.5 mg Daily (N=24)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6) | 1 (2) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 91 (103) | 20 (32) | 13 (13)
Gen disord and admin site conds-Oth spec (General disorders) | 3 (3) | 0 (0) | 0 (0)
Malaise (General disorders) | 5 (5) | 2 (2) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 13 (16) | 4 (7) | 3 (3)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 10 (12) | 3 (5) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 2 (2) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 5 (5) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 93 (108) | 18 (33) | 16 (16)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 9 (10) | 2 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 15 (18) | 4 (7) | 3 (3)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (painful urination) (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 5 (5) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (9) | 4 (5) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 103 (117) | 19 (33) | 15 (15)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT04294225/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT04294225/ICF_000.pdf